CLINICAL TRIAL: NCT02495688
Title: Regional or General Anesthesia for Distal Radius Fracture Surgery in a Day Surgery Setting - A Randomized Clinical Trial
Brief Title: Regional or General Anesthesia for Distal Radius Fracture Surgery in a Day Surgery Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anders Enocson, M.D, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Plx vs GA
Record Dates: First submitted 2015-07-08; First posted 2015-07-13 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Distal Radius Fracture; Postoperative Pain
Keywords: General Anesthesia; Regional Anesthesia
MeSH Terms: conditions — Wrist Fractures; Pain, Postoperative | interventions — Anesthesia, Conduction; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Regional anesthesia (Experimental): Patients are anesthezised with local aneshtetics administered with ultrasound guidance in the nerval plexus of the arm.
  Interventions: Procedure: Regional anesthesia
- General anesthesia (Active Comparator): Patients are anesthezised with general anesthesia and orotrachial airway. Local anesthetics (Chirocaine 5 mg/ml, 10 ml) is administered in the surgical wound during surgery.
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: Regional anesthesia — Standard supraclavicular brachial plexus nerve block. Ultrasound-assisted. By an anesthesiologist. A mix of short- and medium lasting local anesthetics will be used.
  Arms: Regional anesthesia
Procedure: General anesthesia — Standard procedure.
  Arms: General anesthesia

SUMMARY:
The purpose of this study is to compare general and regional anesthesia with regard to postoperative pain in patients who undergo surgery in a day surgery setting due to a displaced distal radius fracture.

DETAILED DESCRIPTION:
We intend to conduct a single-center randomized clinical trial that will enroll 90 patients planned for surgical treatment with a volar plate due to a displaced distal radius fracture in a day surgery setting. Patients who fulfill all of the inclusion criteria and none of the exclusion criteria (see below) will be approached by an MD and/or a RN in the study group on the day of surgery and provided with verbal and written information. If they give their informed written consent to participate in the study they will be randomized to either general or regional anesthesia. The ratio between the study arms will be 1:1 with 45 patients in each group. All patients will receive standard preoperative oral analgesics. Standard procedures for general and regional anesthesia will be used. The regional anesthesia used is supraclavicular brachial nerve block with short- and medium lasting local anesthetics. Patients who receive general anesthesia will be supervised on a postoperative intensive/intermediate care unit until they are stable and have an acceptable pain level before returning to a regular care unit. All patients leave the hospital on the day of surgery. Following standard procedures at our Orthopaedic department all patients will have a non-circular cast for about two weeks for pain-relieve. It will be removed at the standard two week check-up, at which time the sutures are removed, an X-ray is performed and the patients start non-weight bearing mobilization of the wrist.

The primary outcome is total opioid consumption during the first 72 hours postoperatively. It will be measured as the total amount of oral and iv opioids administered in the hospital before discharge as well as oral opioids that the patients consume after discharge. The patients will document their consumption of analgesics in a study diary and for the first three postoperative days report over telephone what they consumed during the previous 24 hours. For details on secondary outcomes see below. The patients will be interviewed over telephone during the first three postoperative days as well as at two weeks. Questions will include grading of pain on a 10 points VAS-scale, grading of postoperative nausea on a 10 points VAS-scale, if they have experienced postoperative vomiting, and if the would recommend the method of anesthesia to a friend or relative. The fractures will be classified by examining X-rays of the fractures before reduction. Postoperative X-rays will be examined and any remaining dislocation will be documented. The patients will fill out an injury-specific (PRWE) and a generic (EQ5D) form for health-related quality of life at the day of surgery (recall for the week before injury) and at 6 months. At 6 months an occupational therapist will perform a test of range of motion (ROM) and grip strength on all patients.

Furthermore, we intend to do an analysis of the resource utilization in the two groups. Time spent in pre-, peri- and postoperative units will be documented for each patient.

All personal data will be handled in a secure way according to ethical and legal regulations.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-74 years planned for surgery with a volar plate due to displaced distal radius fracture.

Exclusion Criteria:

* Dementia,
* alcohol abuse,
* medical condition that interferes with either allocation.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2016-11-12 (Actual); Study Completion 2017-05-16 (Actual)

PRIMARY OUTCOMES:
Postoperative opioid consumption | 72 hours after day care surgery
  The total amount of administered and consumed opioids is calculated for the first 72 hours postoperatively.

SECONDARY OUTCOMES:
Pain | 14 days
  Postoperative pain is recorded on a 10 points VAS-scale directly postoperatively, after two hours, at time of discharge, at 24, 48 and 72 hours, as well as at two weeks postoperatively.
Postoperative Nausea and Vomiting (PONV) | 24 hours
  Nausea is recorded on a 10 points VAS-scale directly postoperatively, after two hours, at time of discharge and at 24 postoperatively. Vomiting during the first 24 hours postoperatively is recorded but not quantified.
PRWE | 6 months
  The injury-specific form, Patient Rated Wrist Evaluation (PRWE), will be filled out by the participants at the day of surgery (recall for the week before injury) as well as at 6 months postoperatively.
EQ5D | 6 months
  The generic form for patient-rated health-related quality of life, EQ5D, will be filled out by the participants at the day of surgery (recall for the week before injury) as well as at 6 months postoperatively.
ROM | 6 months
  Range of motion (ROM) and grip strenght is measured by an unblinded occupational therapist.
X-ray | 14 days
  X-rays of the fracture taken at the emergency department before reduction, as well as at the standard control at the out-patient clinic at 2 weeks after surgery will be examined.

OTHER OUTCOMES:
Resource utilisation | 24 hours
  The utilisation of resources in terms of time in pre-, peri- and postoperative care units will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Anders Enocson, MD, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Södersjukhuset, Stockholm Soder Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Egol KA, Soojian MG, Walsh M, Katz J, Rosenberg AD, Paksima N. Regional anesthesia improves outcome after distal radius fracture fixation over general anesthesia. J Orthop Trauma. 2012 Sep;26(9):545-9. doi: 10.1097/BOT.0b013e318238becb. PMID 22377510